CLINICAL TRIAL: NCT04465123
Title: Furosemide With Early Sequential Nephron Blockade Versus Furosemide Alone in Acute Heart Failure Patients With Furosemide-guided Diuretic Resistance: A Double-blinded, Randomized, Placebo-controlled Study
Brief Title: Early Sequential Nephron Blockade in Acute Heart Failure Patients: A Randomised, Controlled Study
Acronym: NEB-HF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kajohnsak Noppakun, Assistant Professor of Medicine, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MED-2563-07080 (2)
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Acute Heart Failure; Acute Kidney Injury
Keywords: Acute heart failure; Diuretic resistance; Sequential nephron blockade; Diuretic combination
MeSH Terms: conditions — Acute Kidney Injury | interventions — buthiazide, spironolactone drug combination; Spironolactone; Hydrochlorothiazide; Thiazides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furosemide with spironolactone or hydrochlorothiazide (Experimental): IV furosemide dosage will be adjusted according to the protocol as follows. Level 1: previous oral furosemide dose ≤80 mg/day; furosemide 80 mg IV bolus every 6 hours Level 2: previous oral furosemide dose 81-160 mg/day; furosemide 160 mg IV bolus every 6 hours Level 3: previous oral furosemide dose >160 mg/day; furosemide 250 mg IV bolus every 6 hours Furosemide dosage will be adjusted to keep urine output between 3,000 and 5,000 ml/day and >600 ml during 6 hours after furosemide administration.
  If the urine output <3,000 ml/day or <600 ml per 6 hours, furosemide dosage will be increase 1-level up per protocol above.
  If the urine output >5,000 ml/day, furosemide dosage will be reduced 1-level down per protocol above.
  Patients will be received spironolactone or hydrochlorothiazide in combination with intravenous furosemide according to patients' serum potassium levels.
  Interventions: Drug: Spironolactone or hydrochlorothiazide
- Furosemide with placebo (Active Comparator): IV furosemide dosage will be adjusted according to the pre-defined protocol as shown in the experimental group.
  Patients will be received spironolactone placebo or hydrochlorothiazide placebo in combination with intravenous furosemide according to patients' serum potassium levels.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone or hydrochlorothiazide — Patients will be received spironolactone or hydrochlorothiazide in combination with intravenous furosemide according to patients' serum potassium levels.
  If serum potassium levels ≤4 mEq/L, patients will be received spironolactone 100 mg every 12 hour for 72 hours.
  If serum potassium levels >4 mEq/L, patients will be received hydrochlorothiazide 50 mg every 12 hour for 72 hours.
  Other Names: Aldactone; HCTZ; Thiazide
  Arms: Furosemide with spironolactone or hydrochlorothiazide
Drug: Placebo — Patients will be received spironolactone placebo or hydrochlorothiazide placebo in combination with intravenous furosemide according to patients' serum potassium levels.
  If serum potassium levels ≤4 mEq/L, patients will be received spironolactone placebo every 12 hour for 72 hours.
  If serum potassium levels >4 mEq/L, patients will be received hydrochlorothiazide placebo every 12 hour for 72 hours.
  Arms: Furosemide with placebo

SUMMARY:
This study aims to demonstrate the efficacy of sequential nephron blockade by adding hydrochlorothiazide or spironolactone on intravenous furosemide compared to intravenous furosemide alone in the treatments of volume overload in patients with acute heart failure who have diuretic resistance from furosemide stress test.

DETAILED DESCRIPTION:
This study is a randomised, double-blinded, double-dummy, placebo-controlled study to demonstrate the efficacy of oral hydrochlorothiazide or spironolactone in combination with intravenous furosemide compared to intravenous furosemide in combination with placebo. Dosage of intravenous furosemide will be adjusted according to pre-defined protocol. The primary outcome is urine volume during 72 hours after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of acute heart failure which is defined by 2 of the 3 following features: ≥2+ leg edema, jugular venous pressure >10 cm from physical examination or central venous pressure >10 mmHg, and bilateral pulmonary edema or bilateral pleural effusion from chest radiography
* Patients consent to participate into the study

Exclusion Criteria:

* Patients who receive furosemide ≥500 mg/day or hydrochlorothiazide ≥100 mg/day or spironolactone ≥100 mg/day or tolvaptan of any doses
* Patients who have systolic blood pressure <100 mmHg or who need vasoactive drugs inotropic agents (except dobutamine)
* Patients with intravascular volume depletion from clinical evaluation
* Patients with chronic kidney disease stage 5 (estimated glomerular filtration rate <15 ml/min/1.73 m2) or patients who receive maintenance dialysis
* Patients who require renal replacement therapy at the time of admission
* Patients whom diagnosed hypertrophic obstructive cardiomyopathy, severe valvular stenosis or complex congenital heart disease
* Patients with sepsis or systemic infection
* Pregnant women
* Patients who have history of furosemide, spironolactone or hydrochlorothiazide allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Urine volume | 72 hours
  Total urine volume after randomisation

SECONDARY OUTCOMES:
Urine volume | 24 and 48 hours
  Total urine volume after randomization
Body weight | 72 hours after randomisation
  Changes of patient's body weight
Length of hospital admission | During hospital admission period
  Number of days that patients need to stay in the hospital
Furosemide dose | 72 hours after randomisation
  Total dosage of intravenous furosemide
Levels of B-type atrial natriuretic peptide (BNP) | 72 hours and 7 days after randomisation
  levels of pro-BNP
Number of participants with adverse events | During hospital admission
  All adverse events during hospital admission
Dyspnea score assessed by visual analogue scale | At randomization, and 6, 12, 24, 48 and 72 hours after randomization
  The scale is between 0 and 100. The higher scale represents lower level of dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Kajohnsak Noppakun, MD, Principal Investigator — Instructor, Division of Nephrology, Department of Internal Medicine
Locations (1):
- Chiang Mai University Hospital, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No
Request for individual participant data (IPD) has to be submitted to the Institutional Review Board (IRB) of Faculty of Medicine, Chiang Mai University, Chiang Mai, THAILAND.